CLINICAL TRIAL: NCT02469558
Title: Probiotics in Diabesity: A Pilot Study
Acronym: Diabesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 26-464 ex 13/14
Record Dates: First submitted 2015-06-03; First posted 2015-06-11 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- probiotic (Active Comparator): Winclove 851 and 110 consist of 6g of a probiotic mixture containing Bifidobacterium bifidum W23, Bifidobacterium lactis W52, Bifidobacterium lactis W51, Lactobacillus acidophilus W37, Lactobacillus brevis W63, Lactobacillus casei W56, Lactobacillus salivarius W24, Lactococcus lactis W19, Lactococcus lactis W58 at a concentration of 2.5 x 109 cfu/g and 10g of a prebiotic mixture of galacto-oligosaccharides P11 (GOS), Fructo-oligosaccharides P6 (FOS), Konjac glucomannan P13 (E425), Maltodextrin, Calcium carbonate (E170), Natural Elderflower flavouring, Gum Arabic (E414), Zinc citrate 3-hydrate, Vitamin D3 (Cholecalciferol) and Vitamin B2 (Riboflavin) (E101) daily for 6 months
  Interventions: Dietary Supplement: Winclove 851 and 110
- placebo (Placebo Comparator): a similar looking and tasting placebo without bacteria
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Winclove 851 and 110 — prebiotic and probiotic mixture
  Arms: probiotic
Dietary Supplement: Placebo — white powder without pro/probiotic
  Arms: placebo

SUMMARY:
Obesity and type 2 diabetes are a pandemic disease leading to a high morbidity and mortality. Probiotic modulation of gut flora is a possible therapeutic mechanism.

The aim of this study is to investigate and compare thoroughly the effect of a multispecies probiotic on glycaemic control, gut microbiota and gut permeability in patients with metabolic syndrome and diabetes.

DETAILED DESCRIPTION:
Obesity and diabetes probably represent the most challenging threat to public health in the 21st century. The World Health Organization (WHO) predicts that by 2015 approximately 2.3 billion adults will be overweight (BMI 25-29.9 kg/m²), and more than 700 million will be obese (BMI 30 kg/m² or more). In addition, currently 285 million people worldwide suffer from type 2 diabetes (T2DM), and this number is predicted to increase to 439 million by 2030. T2DM raises the risk for cardiovascular morbidity and mortality, as well as eye problems, nerve damage and kidney diseases. Previous studies demonstrated that the impact of diabetes on everyday life and the likelihood of costly and disabling complications can be reduced by more intensive management of glucose, blood pressure and cholesterol. Weight reduction is the most desired but also most difficult to achieve treatment option in obesity, that is able to prevent secondary complications of obesity and T2DM.

Since weight reduction by diet and increased physical activity alone is difficult to achieve in morbidly obese subjects, other, more aggressive approaches, such as bariatric surgery have been invented.

Recent preclinical and clinical studies have indicated an important influence of the intestinal microbiome (gut metagenome) on obesity and associated metabolic disorders (metabolic syndrome, type 2 diabetes, metabolic liver diseases, cardiovascular diseases). For instance, the cecum microbiota of rodents was found to be significantly different in obese than in lean mice. This finding of altered gut microbiota was then confirmed and extended to humans. Additionally, these investigations in humans demonstrated that as obese people lose weight, the composition of microflora shifted, and more closely resembled that of the lean individuals. This suggests that the microflora might be involved in the pathogenesis of obesity, insulin resistance and T2DM by having an impact on gut permeability and chronic inflammation. Probiotic, prebiotic or synbiotic interventions have been shown to be effective in modulating gut permeability and gut microbiota in animals and thereby modulating chronic inflammation and metabolic disorders in animal models. In humans this has not been shown unequivocally so far.

However, it is yet unknown, who will benefit from which intervention and why individuals respond differently to these interventions.

The aim of this study is to investigate and compare thoroughly the effect of a multispecies probiotic on glycaemic control, gut microbiota and gut permeability in patients with metabolic syndrome and diabetes. The investigators aim to access changes in insulin sensitivity, islet function and the secretion of gut hormones. In addition, the investigators will investigate changes in gut microbiota and gut permeability to understand the underlying mechanism. After investigating the mechanism the overarching aim is to identify biomarkers, which would allow better prediction of treatment success. In future this would allow tailoring obesity and diabetes treatment in order to give every patient the optimal treatment at lowest costs.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Age above 18 years
* Type 2 diabetes
* BMI 30-40 kg/m²
* HbA1c ≥ 6.5% (48 mmol/mol)
* Stable diabetes therapy over 6 months
* Person commits to the need for long-term follow-up

Exclusion Criteria:

* Type 1 diabetes mellitus
* Maturity Onset Diabetes of the Young (MODY)
* Secondary diabetes due to a specific disease or glucocorticoid therapy
* Pregnancy
* Hypothalamic cause of obesity, Cushing syndrome
* Major psychiatric diseases including diagnosed eating disorders, history of drug or alcohol abuse
* History of bariatric surgery
* Use of probiotics (other than the study product)
* Antibiotic therapy within the last 4 weeks before inclusion
* Inflammatory bowel disease
* Pancreatitis
* Chronic non-steroidal anti-inflammatory drug (NSAID) treatment
* glucagon-like peptide-1 receptor agonist therapy or acarbose therapy
* Recent (less than 12 weeks) acute myocardial infarction or decompensated heart failure
* Recent (less than 12 weeks) stroke
* Known malignancy or any other condition or circumstance, which, in the opinion of the investigator, would affect the patient's ability to participate in the protocol

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-09; Primary Completion 2018-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
insulin sensitivity | 12 months
  meal tolerance test

OTHER OUTCOMES:
gut microbiota composition | 12 months
  next generation sequencing
gut permeability | 12 months
  enzyme linked immunosorbent assay
endotoxin | 12 months
  limulus amoebocyte assay
neutrophil function | 12 months
  flow cytometry
beta cell function | 12 months
  meal tolerance test
Quality of Life | 12 months
  quality of life questionnaire (short form 36, Subscores for 8 domains)

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Stadlbauer-Köllner, MD, Principal Investigator — Medical University of Graz; Harald Sourij, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Department of Internal Medicine, Graz, Austria